CLINICAL TRIAL: NCT04887766
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Assessing the Effect of GS300 on Nonalcoholic Fatty Liver Disease
Brief Title: Study on GS300 on NAFLD
Acronym: REVERT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gelesis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-300-001
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Nonalcoholic Fatty Liver; Weight Loss
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Weight Loss

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): GS300: Three (3) GS300 capsules [approximately 0.65 grams (g)] two (2) times per day ingested 10 minutes (min) before meals (i.e., lunch and dinner) - total of 3.9 g per day
  Interventions: Device: GS300
- Placebo (Placebo Comparator): Placebo: Three (3) placebo capsules two (2) times per day 10 min before meals (i.e., lunch and dinner)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: GS300 — Gelesis300 hydrogel in gelatin capsules
  Arms: Active
Device: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
To determine the efficacy of GS300 when administered for 24 weeks in patients with Nonalcoholic Fatty Liver Disease (NAFLD).

DETAILED DESCRIPTION:
This is a multicenter, randomized, placebo-controlled, double-blinded, parallel-group study. Patients will be randomized 1:1 to receive either GS300 or placebo. The study includes an up to 6 weeks screening period, a 24-week treatment period, and a 1-week follow-up period.

Approximately 250 patients (125 patients per arm) will be enrolled (at least 40% from each gender and at least 40% from US and 40% from Europe).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 22 years and ≤ 65 years
2. Body Mass Index (BMI) ≥ 27 and ≤ 40 kilogram (kg)/meter2 (m2)
3. Negative for Hepatitis B, C and Human Immunodeficiency Virus (HIV) within 6 months of screening [HbsAg negative and Hepatitis C Virus (HCV) RNA negative; subjects treated and cured of HCV must have completed treatment and tested negative for HCV at least 2 years prior to study enrollment]
4. Fibroscan CAP score > 300 decibels (dB)/m
5. Stable body weight defined as less than 5% change in body weight in the 3 months prior to screening (per patient report)
6. Approximately 250 patients (approximately 125 patients per treatment arm)

   1. Prediabetes i) Untreated prediabetic patients with FPG ≥ 100 mg/ dL (≥ 5.6 mmol/L) and < 126 mg/dL (< 7.0 mmol/L) at both Screening Visits with HbA1c ≤ 6.4% (≤ 46 mmol/mol) - if only one value is within this range, the other value should not be ≥ 126 mg/dL (≥ 7.0 mmol/L) and HbA1c should be ≥ 5.7% (≥ 39 mmol/mol) and ≤ 6.4% (≤ 46 mmol/mol) ii) Drug-treated (metformin) prediabetic patients with FPG ≥ 70 mg/dL (≥ 3.9 mmol/L) and < 126 mg/dL (< 7.0 mmol/L) at both Screening Visits
   2. Type 2 Diabetes i) Untreated type 2 diabetic patients with FPG ≤ 200 mg/dL (≤ 11.2 mmol/L) at both Screening Visits and either FPG ≥ 126 mg/dL (≥ 7.0 mmol/L) at both Screening Visits or FPG < 126 mg/dL (< 7.0 mmol/L) at one or both Screening Visits with HbA1c ≥ 6.5% (≥ 48 mmol/mol) ii) Drug-treated [metformin and/or dipeptidyl peptidase-4 (DPP-4) inhibitors, and/or insulin] type 2 diabetic patients with FPG ≥ 70 mg/dL (≥ 3.9 mmol/L) and ≤ 270 mg/dL (≤ 15.1 mmol/L) at both Screening Visits Note, approximately 10% to 20% of enrolled Type 2 diabetic patients will be on insulin therapy
   3. Normoglycemia (up to approximately 10% of patients) Normoglycemic patients with FPG ≥ 70 mg/dL (≥ 3.9 mmol/L) and < 100 mg/ dL (< 5.6 mmol/L) at both Screening Visits with HbA1c < 5.7% (< 39 mmol/mol) and HOMA-IR ≥ 3.0
7. MRI PDFF ≥ 10%
8. Willing to sign the ICF prior to any study related procedures

Exclusion Criteria:

1. Self-reported alcohol intake > 20 gram (g)/day for women and > 30 g/day for men (on average per day) as per medical history
2. Alcohol Use Disorders Identification Test (AUDIT) questionnaire: AUDIT-C score of ≥ 4 in men and ≥ 3 in women will be followed by a full AUDIT questionnaire by interview with patients excluded for score ≥ 8
3. Prior liver transplant
4. Liver cirrhosis as evidenced by any of the following:

   * Serum albumin < 3.5 g/dL (0.53 mmol/L)
   * INR > 1.3 (unless due to anticoagulant therapy)
   * AST/ALT ratio ≥ 2
   * Direct bilirubin > 0.3 mg/dL (5.13 micromol (micromol)/L)
   * Platelet count < 150,000/microL
5. History or evidence of other chronic liver diseases, including, but not limited to the following:

   * Current active autoimmune hepatitis
   * Primary biliary cholangitis (PBC)
   * Primary sclerosing cholangitis
   * Wilson's disease
   * Alpha-1-antitrypsin (A1AT) deficiency
   * Hemochromatosis
   * Drug-induced liver disease, as defined on the basis of typical exposure and history
   * Bile duct obstruction
   * Suspected or proven liver cancer
   * History of hepatic encephalopathy
   * Portal hypertension (esophageal varices, ascites, splenomegaly)
6. History of gastric surgery (up to 10% patients with history of gastric bypass or sleeve gastrectomy may be enrolled if the surgery occurred more than 6 months prior to enrollment and patients had a weight change < 5% during the 3 months prior to enrollment)
7. Angina, coronary bypass, or myocardial infarction within 6 months prior to Screening Visit
8. Inflammatory bowel disease, celiac disease, or other significant gastrointestinal disease - for example, a history of bowel obstruction without surgical correction (patients with irritable bowel syndrome may be enrolled)
9. Pregnancy
10. Absence of medically approved contraceptive methods in females of childbearing potential (e.g., hysterectomy, oral contraceptives, non-oral contraceptive medications or intrauterine device combined with a barrier method, two combined barrier methods such as diaphragm and condom or spermicide, or condom and spermicide; bilateral tubal ligation and vasectomy are not acceptable methods)
11. Type 1 Diabetes
12. HbA1c > 8.5% (> 69 mmol/mol)
13. Serum LDL-C ≥ 160 mg/dL (≥ 4.15 mmol/L)
14. Serum triglycerides ≥ 350 mg/dL (≥ 3.96 mmol/L)
15. Use of any medications for the treatment of diabetes within 3 months prior to enrollment. Note, metformin, DPP-4 inhibitors, and insulin at a stable dose over the last 3 months are allowed. Insulin dose variance of 20% (decrease or increase) is allowed.
16. Any change in standard of care or background therapy for liver disease or other ongoing chronic conditions within 3 months prior to enrollment, including changes in the following:

    * Antidiabetic medications (metformin, DPP-4 inhibitors, insulin)
    * Thyroid hormones
    * Medications treating depression
    * Medications treating dyslipidemia
    * Medications treating hypertension
    * Vitamin E
17. Regular/daily use of any of the following within 3 months prior to enrollment or anticipated regular/daily use during the study period:

    * High dose nonsteroidal anti-inflammatory drugs (NSAIDS) (equivalent of > 3,200 mg/day ibuprofen)
    * Systemic corticosteroids, anabolic steroids
    * Methotrexate, amiodarone, tamoxifen, tetracyclines, estrogens at doses greater than those used for hormone replacement, valproic acid
    * Probiotic supplements (yogurt is allowed)
    * Addictive, non-prescribed medications including amphetamines, barbiturates, cocaine, opiates, methadone and phencyclidine as per medical history or regular daily use of cannabinoids
18. Use of any anti-obesity medications (including herbal preparations) within 2 months prior to enrollment or any anticipated use during the study period
19. History of allergic reaction to carboxymethylcellulose (CMC), citric acid, sodium stearyl fumarate, raw cane sugar, gelatin, or titanium dioxide
20. Currently enrolled in another investigational device or drug study, or less than 3 months since ending another investigational device or drug study(s), or receiving other investigational treatment(s)
21. Any disease or condition that, in the opinion of the investigator or Sponsor, would interfere with study participation

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss ≥ 5% | 24 Weeks
  Proportion of patients with weight loss ≥ 5% at Week 24.
Placebo-adjusted percent change in weight from Baseline to Week 24 | 24 Weeks
  Placebo-adjusted percent change in weight from Baseline to Week 24.
Relative reduction in liver fat | 24 Weeks
  Relative reduction in liver fat from Baseline to Week 24, as measured by hepatic Magnetic Resonance Imaging Proton Density Fat Fraction (MRI PDFF).

SECONDARY OUTCOMES:
Weight loss ≥ 7.5% | 24 Weeks
  To assess reduction in weight (≥ 7.5%) in patients with NAFLD treated with GS300 or placebo.
Weight loss ≥ 10% | 24 Weeks
  To assess reduction in weight (≥ 10%) in patients with NAFLD treated with GS300 or placebo.
To evaluate the percentage of patients with ≥ 30% relative reduction in liver fat | 24 Weeks
  To evaluate the percentage of patients with ≥ 30% relative reduction in liver fat in patients treated with GS300 or placebo.
To assess placebo-adjusted waist circumference reduction | 24 Weeks
  To assess placebo-adjusted waist circumference reduction after 24 weeks of treatment with GS300 or placebo.
To assess the impact of GS300 on glycemic control in patients with NAFLD | 24 Weeks
  To assess the impact of GS300 on glycemic control in patients with NAFLD treated with GS300 or placebo.
To assess the impact of GS300 on liver enzymes in patients with NAFLD | 24 Weeks
  To assess the impact of GS300 on liver enzymes in patients with NAFLD treated with GS300 or placebo.

OTHER OUTCOMES:
Intestinal Permeability | 24 Weeks
  Intestinal permeability - Urine test (sub-population of 50 patients at selected sites).
Vitamin Levels | 24 Weeks
  Serum/plasma vitamin levels (sub-population at selected sites).
Gut Peptides | 24 Weeks
  Glucagon-like Peptide-1 (GLP-1), Glucagon-like Peptide-2 (GLP-2), Gastric Inhibitory Polypeptide (GIP), ghrelin, somatostatin, Cholecystokinin (CCK), Peptide YY (PYY).

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Heshmati, MD, Study Director — Gelesis, Inc.